CLINICAL TRIAL: NCT00506350
Title: Evaluate the Reactogenicity & Immunogenicity of 1 or 2 Booster Administrations of an Influenza Pandemic Candidate Vaccine (GSK1562902A) in Primed Adults Aged Between 19 & 61 Years
Brief Title: Evaluate Reactogenicity & Immunogenicity of an Influenza Pandemic Candidate Vaccine (GSK1562902A) in Primed Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109817
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Results first posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Influenza
MeSH Terms: conditions — Influenza, Human

ARMS (9):
- GSK1562902A non-AD F1 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of a non-adjuvanted (non-AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 1 (F1) in study 106750 (NCT00309634) receiving 2 doses of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, one at Day 0 and one at Day 21, administrated intramuscularly (IM) in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 2 doses
- GSK1562902A non-AD F2 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of a non-adjuvanted (non-AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 2 (F2) in study 106750 (NCT00309634) receiving 2 doses of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, one at Day 0 and one at Day 21, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 2 doses
- GSK1562902A non-AD F3 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of a non-adjuvanted (non-AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 3 (F3) in study 106750 (NCT00309634) receiving 2 doses of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, one at Day 0 and one at Day 21, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 2 doses
- GSK1562902A non-AD F4 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of a non-adjuvanted (non-AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 4 (F4) in study 106750 (NCT00309634) receiving 2 doses of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, one at Day 0 and one at Day 21, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 2 doses
- GSK1562902A AD F1 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of an adjuvanted (AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation1 (F1) in study 106750 (NCT00309634) received 1 dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study at Day 0, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 1 dose
- GSK1562902A AD F2 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of an adjuvanted (AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 2 (F2) in study 106750 (NCT00309634) received 1 dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study at Day 0, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 1 dose
- GSK1562902A AD F3 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of an adjuvanted (AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 3 (F3)in study 106750 (NCT00309634) received 1 dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study at Day 0, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 1 dose
- GSK1562902A AD Approved F4 Primed Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of approved Formulation (F) of adjuvanted (AD) H5N1 vaccine (A/Vietnam/1194/04 strain) in study 106750 (NCT00309634) received 1 dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study at Day 0, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 1 dose
- Control Group (Experimental): Healthy male or female adults, between and including 19 to 61 years of age, unprimed receiving 2 doses of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study, one at Day 0 and one at Day 21, administrated IM in the deltoid region of the non-dominant arm.
  Interventions: Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 2 doses

INTERVENTIONS:
Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 1 dose — A single dose of Pandemic influenza candidate vaccine (GSK1562902A) administered intramuscularly in the deltoid region of the non-dominant arm at Day 0.
  Arms: GSK1562902A AD Approved F4 Primed Group; GSK1562902A AD F1 Primed Group; GSK1562902A AD F2 Primed Group; GSK1562902A AD F3 Primed Group
Biological: Pandemic influenza candidate vaccine (GSK1562902A) - 2 doses — Two doses of Pandemic influenza candidate vaccine (GSK1562902A) administered intramuscularly in the deltoid region of the non-dominant arm at Day 0 and Day 21.
  Arms: Control Group; GSK1562902A non-AD F1 Primed Group; GSK1562902A non-AD F2 Primed Group; GSK1562902A non-AD F3 Primed Group; GSK1562902A non-AD F4 Primed Group

SUMMARY:
The present study is designed to evaluate the reactogenicity and immunogenicity of one or two booster administrations of an influenza pandemic candidate vaccine (GSK1562902A) in adults aged between 19 and 61 years, previously vaccinated with 2 doses of a pandemic candidate vaccine. Fifty new subjects who did not participate in a primary study (106750, NCT00309634) will be recruited. This protocol posting deals with objectives & outcome measures of the booster phase. The objectives & outcome measures of the primary phase are presented in a separate protocol posting (NCT00309634)

DETAILED DESCRIPTION:
The present study is designed to evaluate the reactogenicity and immunogenicity of one or two booster administrations of an influenza pandemic candidate vaccine (GSK1562902A) in adults aged between 19 and 61 years, previously vaccinated with 2 doses of a pandemic candidate vaccine. The persistence of antibodies will be analysed at 6, 12, 18 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes can and will comply with the requirements of the protocol should be enrolled in the study.
* For previously primed subjects: participation in the primary study (NCT00309634).
* For unprimed subjects: male or female between and including, 19 and 61 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* If the subject is female, she must be of non-childbearing potential or if she is of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* For unprimed subjects who did not participate in the primary study (NCT00309634): Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a licenced vaccine not foreseen by the study protocol within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) of the first dose of vaccine(s).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Applicable for control group only: previous vaccination with a pandemic candidate vaccine or a vaccine containing the investigational vaccine adjuvant.
* History of hypersensitivity to vaccines.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required).
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccine(s).
* Major congenital defects or serious chronic illness.
* History of any neurological disorders or seizures.
* Acute disease at the time of enrolment.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Serious chronic disease including any medically significant chronic pulmonary, cardiovascular, renal, neurological, psychiatric or metabolic disorder, as determined by medical history and physical examination.
* Any condition which, in the opinion of the investigator, prevents the subject from participation in the study.
* Lactating female.
* History of chronic alcohol consumption and/or drug abuse

Ages: 19 Years to 61 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2007-08-01 (Actual); Primary Completion 2009-10-12 (Actual); Study Completion 2009-10-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109817 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Groups:
- GSK1562902A AD F3 Primed Group: Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of an adjuvanted (AD) investigational H5N1 vaccine (A/Vietnam/1194/04 strain) Formulation 3 (F3) in study 106750 (NCT00309634) received 1 dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study at Day 0, administrated IM in the deltoid region of the non-dominant arm.
- GSK1562902A AD Approved F Primed Group: Healthy male or female adults, between and including 19 to 61 years of age, primed with 2 doses of approved Formulation (F) of adjuvanted (AD) H5N1 vaccine (A/Vietnam/1194/04 strain) in study 106750 (NCT00309634) received 1 dose of Pandemic influenza candidate vaccine (GSK1562902A) in this booster study at Day 0, administrated IM in the deltoid region of the non-dominant arm.
Period: Overall Study
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Started | 36 | 40 | 37 | 36 | 50 | 40 | 35 | 41 | 35
Completed | 33 | 37 | 31 | 34 | 40 | 38 | 33 | 36 | 30
Not Completed | 3 | 3 | 6 | 2 | 10 | 2 | 2 | 5 | 5
Not completed — Serious Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 4 | 1 | 1 | 2 | 0
Not completed — Lost to Follow-up | 1 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 2
Not completed — Medical Reason | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 3 | 0 | 3 | 0 | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group | Total
Number analyzed (Participants) | 36 | 40 | 37 | 36 | 50 | 40 | 35 | 41 | 35 | 350
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.3 (12.80) | 36.3 (12.36) | 36.8 (12.87) | 39.5 (13.27) | 32.1 (9.96) | 38.5 (13.43) | 38.3 (14.61) | 34.8 (14.57) | 35.9 (12.78) | 36.32 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 16 | 21 | 34 | 27 | 18 | 23 | 18 | 194
  Male | 18 | 21 | 21 | 15 | 16 | 13 | 17 | 18 | 17 | 156
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White - Arabic / North African heritage | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Race: White - Caucasian / European heritage | 36 | 38 | 37 | 36 | 48 | 40 | 34 | 41 | 35 | 345
  Race: Other | 0 | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Titers for Serum H5N1 Haemagglutinin Inhibition (HI) Antibodies Against the A/Indonesia/05/2005 Strain
Description: Titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:10. The flu strain assessed was A/Indonesia/05/2005.
Time Frame: At Day 0
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 39 | 33 | 38 | 32
Titers | 5.1 [4.9 to 5.3] | 5.6 [4.8 to 6.5] | 5.3 [4.9 to 5.8] | 5.2 [4.8 to 5.5]

2. Primary Outcome: Titers for Serum H5N1 Haemagglutinin Inhibition (HI) Antibodies Against the A/Indonesia/05/2005 Strain
Description: as for outcome 1
Time Frame: At Day 21
Population: The analysis was performed on the ATP cohort for immunogenicity, which included all evaluable subjects for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 39 | 33 | 38 | 33
Titers | 406.8 [225.9 to 732.7] | 429.5 [281.2 to 655.9] | 208.4 [126.3 to 343.9] | 347.9 [213.6 to 566.8]

3. Primary Outcome: Number of Seroconverted Subjects for H5N1 HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroconversion rate for HI antibody response was defined as the percentage of vaccines who have either a pre-vaccination titer < 1:10 and a post-vaccination titer ≥ 1:40 or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 39 | 33 | 38 | 32
Participants | 36 | 33 | 34 | 31

4. Primary Outcome: Seroconversion Factor (SCF) for H5N1 HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroconversion factor (SCF) was defined as the fold increase in H5N1 HI antibody GMTs post-vaccination compared to Day 0. The flu strain assessed was A/Indonesia/05/2005.
Time Frame: At Day 21
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 39 | 33 | 38 | 32
Fold increase | 79.9 [44.5 to 143.6] | 76.5 [50.7 to 115.6] | 39.1 [24.2 to 63.1] | 76.9 [51.5 to 115.0]

5. Primary Outcome: Number of Seroprotected Subjects for H5N1 HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer equal to or above (≥) 1:40. The flu strain assessed was A/Indonesia/05/2005.
Time Frame: At Day 0
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 39 | 33 | 38 | 32
Participants | 0 | 1 | 0 | 0

6. Primary Outcome: Number of Seroprotected Subjects for H5N1 HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: as for outcome 5
Time Frame: At Day 21
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 39 | 33 | 38 | 33
Participants | 36 | 33 | 34 | 31

7. Primary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms
Description: Assessed solicited local symptoms were ecchymosis, induration, pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 ecchymosis/induration/redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site. No subject from GSK1562902A AD F1 Primed Group has received Dose 2.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available and who had their symptom sheets filled in.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 36 | 40 | 36 | 36 | 50 | 40 | 35 | 41 | 35
Participants
  Any Ecchymosis, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Ecchymosis, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration, Dose 1 | 5 | 1 | 3 | 2 | 2 | 2 | 3 | 3 | 4
  Grade 3 Induration, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Dose 1 | 33 | 35 | 32 | 34 | 45 | 38 | 34 | 39 | 31
  Grade 3 Pain, Dose 1 | 2 | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 0
  Any Redness, Dose 1 | 0 | 1 | 0 | 0 | 1 | 1 | 3 | 1 | 1
  Grade 3 Redness, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Dose 1 | 4 | 2 | 4 | 4 | 3 | 2 | 2 | 3 | 2
  Grade 3 Swelling, Dose 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any Ecchymosis, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Ecchymosis, Dose 2 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Grade 3 Ecchymosis, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Ecchymosis, Dose 2 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Any Induration, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Induration, Dose 2 | 1 | 5 | 3 | 1 | 4 |  | 1 | 0 | 0
  Grade 3 Induration, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Induration, Dose 2 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Pain, Dose 2 | 28 | 30 | 24 | 28 | 42 |  | 1 | 1 | 1
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Pain, Dose 2 | 0 | 0 | 0 | 0 | 2 |  | 0 | 0 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Redness, Dose 2 | 0 | 1 | 0 | 0 | 2 |  | 1 | 0 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Redness, Dose 2 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Swelling, Dose 2 | 3 | 0 | 2 | 5 | 5 |  | 1 | 0 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Swelling, Dose 2 | 0 | 0 | 0 | 0 | 1 |  | 0 | 0 | 0
  Any Ecchymosis, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Ecchymosis, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration, Across doses | 6 | 5 | 5 | 2 | 6 | 2 | 4 | 3 | 4
  Grade 3 Induration, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain, Across doses | 34 | 36 | 32 | 35 | 47 | 38 | 34 | 39 | 31
  Grade 3 Pain, Across doses | 2 | 0 | 0 | 2 | 3 | 1 | 1 | 1 | 0
  Any Redness, Across doses | 0 | 1 | 0 | 0 | 3 | 1 | 4 | 1 | 1
  Grade 3 Redness, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling, Across doses | 5 | 2 | 5 | 6 | 6 | 2 | 3 | 3 | 2
  Grade 3 Swelling, Across doses | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms
Description: Assessed solicited general symptoms were arthralgia, fatigue, headache, myalgia, shivering, sweating and fever [defined as axillary temperature equal to or above (≥) 38 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever ≥ 39.0 °C. Related = symptom assessed by the investigator as causally related to the study vaccination. No subject from GSK1562902A AD F1 Primed Group has received Dose 2.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each dose and across doses
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 36 | 40 | 36 | 36 | 50 | 40 | 35 | 41 | 35
Participants
  Any Arthralgia, Dose 1 | 5 | 7 | 2 | 5 | 9 | 6 | 5 | 5 | 5
  Grade 3 Arthralgia, Dose 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Related Arthralgia, Dose 1 | 4 | 5 | 2 | 5 | 7 | 5 | 5 | 5 | 4
  Any Fatigue, Dose 1 | 12 | 15 | 15 | 15 | 24 | 15 | 10 | 18 | 13
  Grade 3 Fatigue, Dose 1 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0
  Related Fatigue, Dose 1 | 10 | 12 | 15 | 13 | 22 | 15 | 9 | 17 | 12
  Any Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Dose 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache, Dose 1 | 14 | 15 | 12 | 11 | 14 | 19 | 10 | 11 | 9
  Grade 3 Headache, Dose 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 0
  Related Headache, Dose 1 | 11 | 11 | 11 | 10 | 11 | 16 | 9 | 10 | 8
  Any Myalgia, Dose 1 | 12 | 17 | 14 | 12 | 18 | 12 | 12 | 11 | 10
  Grade 3 Myalgia, Dose 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
  Related Myalgia, Dose 1 | 12 | 15 | 14 | 10 | 17 | 11 | 11 | 9 | 9
  Any Shivering, Dose 1 | 4 | 1 | 1 | 5 | 7 | 9 | 6 | 6 | 3
  Grade 3 Shivering, Dose 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Related Shivering, Dose 1 | 4 | 1 | 1 | 4 | 6 | 9 | 6 | 5 | 3
  Any Sweating, Dose 1 | 2 | 4 | 6 | 3 | 10 | 5 | 6 | 4 | 3
  Grade 3 Sweating, Dose 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Related Sweating, Dose 1 | 2 | 2 | 6 | 2 | 6 | 5 | 6 | 3 | 3
  Any Arthralgia, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Arthralgia, Dose 2 | 9 | 4 | 5 | 6 | 10 |  | 0 | 0 | 0
  Grade 3 Arthralgia, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Arthralgia, Dose 2 | 1 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Related Arthralgia, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Arthralgia, Dose 2 | 6 | 4 | 5 | 6 | 10 |  | 0 | 0 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Fatigue, Dose 2 | 13 | 12 | 9 | 13 | 25 |  | 0 | 1 | 0
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Fatigue, Dose 2 | 1 | 0 | 0 | 0 | 3 |  | 0 | 0 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Fatigue, Dose 2 | 12 | 10 | 6 | 13 | 24 |  | 0 | 1 | 0
  Any Fever, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Fever, Dose 2 | 1 | 1 | 0 | 0 | 4 |  | 0 | 0 | 0
  Grade 3 Fever, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Fever, Dose 2 | 0 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Related Fever, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Fever, Dose 2 | 1 | 1 | 0 | 0 | 4 |  | 0 | 0 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Headache, Dose 2 | 14 | 10 | 12 | 9 | 23 |  | 0 | 1 | 0
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Headache, Dose 2 | 0 | 0 | 0 | 0 | 3 |  | 0 | 0 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Headache, Dose 2 | 12 | 9 | 8 | 9 | 19 |  | 0 | 1 | 0
  Any Myalgia, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Myalgia, Dose 2 | 11 | 9 | 9 | 7 | 24 |  | 0 | 1 | 0
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Myalgia, Dose 2 | 1 | 0 | 0 | 0 | 0 |  | 0 | 0 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Myalgia, Dose 2 | 11 | 8 | 9 | 6 | 22 |  | 0 | 1 | 0
  Any Shivering, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Shivering, Dose 2 | 7 | 3 | 4 | 3 | 14 |  | 0 | 1 | 0
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Shivering, Dose 2 | 0 | 0 | 0 | 0 | 1 |  | 0 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Shivering, Dose 2 | 6 | 3 | 4 | 3 | 14 |  | 0 | 1 | 0
  Any Sweating, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Any Sweating, Dose 2 | 7 | 2 | 3 | 2 | 10 |  | 0 | 1 | 0
  Grade 3 Sweating, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Grade 3 Sweating, Dose 2 | 0 | 0 | 0 | 0 | 1 |  | 0 | 0 | 0
  Related Sweating, Dose 2: number analyzed (Participants) | 35 | 40 | 36 | 33 | 49 | 0 | 1 | 1 | 1
  Related Sweating, Dose 2 | 5 | 2 | 3 | 2 | 10 |  | 0 | 1 | 0
  Any Arthralgia, Across doses | 13 | 8 | 6 | 10 | 14 | 6 | 5 | 5 | 5
  Grade 3 Arthralgia, Across doses | 2 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0
  Related Arthralgia, Across doses | 10 | 6 | 6 | 10 | 13 | 5 | 5 | 5 | 4
  Any Fatigue, Across doses | 20 | 21 | 17 | 20 | 30 | 15 | 10 | 18 | 13
  Grade 3 Fatigue, Across doses | 2 | 0 | 0 | 0 | 5 | 1 | 0 | 1 | 0
  Related Fatigue, Across doses | 17 | 18 | 17 | 20 | 29 | 15 | 9 | 17 | 12
  Any Fever, Across doses | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
  Grade 3 Fever, Across doses | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Related Fever, Across doses | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
  Any Headache, Across doses | 20 | 17 | 17 | 14 | 28 | 19 | 10 | 11 | 9
  Grade 3 Headache, Across doses | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 1 | 0
  Related Headache, Across doses | 18 | 16 | 14 | 14 | 22 | 16 | 9 | 10 | 8
  Any Myalgia, Across doses | 17 | 20 | 15 | 15 | 30 | 12 | 12 | 11 | 10
  Grade 3 Myalgia, Across doses | 3 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
  Related Myalgia, Across doses | 17 | 18 | 15 | 14 | 28 | 11 | 11 | 9 | 9
  Any Shivering, Across doses | 10 | 3 | 4 | 7 | 20 | 9 | 6 | 6 | 3
  Grade 3 Shivering, Across doses | 1 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0
  Related Shivering, Across doses | 9 | 3 | 4 | 7 | 19 | 9 | 6 | 5 | 3
  Any Sweating, Across doses | 9 | 4 | 6 | 5 | 13 | 5 | 6 | 4 | 3
  Grade 3 Sweating, Across doses | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
  Related Sweating, Across doses | 7 | 3 | 6 | 4 | 12 | 5 | 6 | 3 | 3

9. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevented normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day (Days 0-20) follow-up period after the first vaccination and 30-day (Days 0-29) follow-up period after the second vaccination
Population: The analysis was performed on the Total Vaccinated cohort, which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group
Number analyzed (Participants) | 36 | 40 | 37 | 36 | 50
Participants
  Any AE(s) | 22 | 24 | 21 | 26 | 33
  Grade 3 AE(s) | 2 | 4 | 1 | 3 | 6
  Related AE(s) | 4 | 1 | 4 | 1 | 8

10. Primary Outcome: Number of Subjects With Any, Grade 3 and Related Unsolicited Adverse Events (AEs)
Description: as for outcome 9
Time Frame: During the 30-day (Days 0-29) follow-up period after the first vaccination
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 40 | 35 | 41 | 35
Participants
  Any AE(s) | 13 | 17 | 17 | 17
  Grade 3 AE(s) | 3 | 2 | 5 | 2
  Related AE(s) | 5 | 4 | 4 | 4

11. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life-threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: During the entire study period (From Day 0 up to Month 24)
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 36 | 40 | 37 | 36 | 50 | 40 | 35 | 41 | 35
Participants
  Day 0 - Month 6 | 1 | 1 | 1 | 0 | 3 | 1 | 0 | 1 | 0
  Month 6 - Month 12 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Month 12 - Month 18 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2
  Month 18 - Month 24 | 1 | 1 | 1 | 0 | 0 | 1 | 0 | 1 | 2

12. Secondary Outcome: Titers for Serum Neutralizing HI Antibodies Against A/Indonesia/05/2005 Strain
Description: Titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:28. The flu strain assessed was A/Indonesia/05/2005. No subject from GSK1562902A AD F1 Primed Group has received a second vaccination.
Time Frame: At Days 0, 21 (post-vaccination one) and 42 (post-vaccination two)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A AD F1 Primed Group | Control Group
Number analyzed (Participants) | 34 | 38 | 49
Titers
  A/Indonesia/05/2005, Day 0 | 47.0 [34.2 to 64.6] | 157.8 [130.3 to 191.2] | 19.9 [15.7 to 25.2]
  A/Indonesia/05/2005, Day 21: number analyzed (Participants) | 34 | 0 | 49
  A/Indonesia/05/2005, Day 21 | 692.4 [476.7 to 1005.7] |  | 307.3 [262.5 to 359.8]
  A/Indonesia/05/2005, Day 42 | 933.1 [653.7 to 1331.9] | 3708.9 [2458.6 to 5594.9] | 1606.4 [1282.7 to 2011.8]

13. Secondary Outcome: Titers for Serum Neutralizing HI Antibodies Against A/Indonesia/05/2005 Stain
Description: Titers were presented as geometric mean titers (GMTs). The reference seropositivity cut-off value was equal to or above (≥) 1:28. The flu strain assessed was A/Indonesia/05/2005.
Time Frame: At Months 6, 12, 18 and 24
Population: The analysis was performed on the ATP cohort for persistence, which included all subjects who had serologic results available at the antibody persistence time-point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A Non-AD F1 Primed Group | Control Group
Number analyzed (Participants) | 37 | 35 | 46
Titers
  A/Indonesia/05/2005, Month 6 | 1422.2 [916.8 to 2206.2] | 502.3 [349.2 to 722.5] | 751.3 [611.4 to 923.3]
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 37 | 32 | 44
  A/Indonesia/05/2005, Month 12 | 557.6 [354.0 to 878.4] | 180.7 [121.3 to 269.2] | 274.4 [215.7 to 349.1]
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 34 | 31 | 37
  A/Indonesia/05/2005, Month 18 | 767.5 [494.8 to 1190.6] | 278.5 [173.7 to 446.5] | 569.9 [442.9 to 733.4]
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 34 | 30 | 32
  A/Indonesia/05/2005, Month 24 | 503.2 [338.3 to 748.4] | 201.6 [143.2 to 283.8] | 295.4 [237.8 to 367.0]

14. Secondary Outcome: Titers for Serum H5N1 Haemaglutinin-inhibition (HI) Antibodies Against the A/Indonesia/05/2005 Strain
Description: as for outcome 1
Time Frame: At Days 0, 7, 14, 21, 28, 35 and 42
Population: The analysis was performed on the ATP cohort for immunogenicity, whiich included all evaluable subjects for whom immunogenicity data and assay results for antibodies against at least one study vaccine antigen component after vaccination were available.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group
Number analyzed (Participants) | 34 | 38 | 33 | 28 | 49
Titers
  A/Indonesia/05/2005, Day 0 | 5.1 [4.9 to 5.3] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0] | 5.0 [5.0 to 5.0]
  A/Indonesia/05/2005, Day 7 | 22.1 [11.7 to 41.8] | 25.3 [14.5 to 44.4] | 27.7 [16.1 to 47.6] | 37.6 [19.3 to 73.4] | 5.0 [5.0 to 5.0]
  A/Indonesia/05/2005, Day 14: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 14 | 46.6 [24.0 to 90.7] | 66.1 [39.7 to 109.9] | 49.1 [25.7 to 93.8] | 71.5 [39.0 to 131.2] | 13.7 [9.6 to 19.5]
  A/Indonesia/05/2005, Day 21: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 21 | 38.0 [20.4 to 70.6] | 57.6 [36.9 to 90.0] | 42.2 [23.0 to 77.4] | 77.1 [45.1 to 131.7] | 31.0 [20.8 to 46.3]
  A/Indonesia/05/2005, Day 28: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 28 | 48.1 [26.1 to 88.7] | 79.3 [52.7 to 119.3] | 56.0 [31.2 to 100.4] | 128.0 [81.8 to 200.4] | 543.9 [423.3 to 698.8]
  A/Indonesia/05/2005, Day 35: number analyzed (Participants) | 33 | 36 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 35 | 56.0 [28.6 to 109.8] | 119.9 [77.5 to 185.5] | 65.8 [36.1 to 120.2] | 160.0 [100.8 to 254.2] | 563.6 [438.5 to 724.4]
  A/Indonesia/05/2005, Day 42: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 42 | 54.3 [27.9 to 105.8] | 116.3 [77.2 to 175.4] | 63.7 [34.5 to 117.9] | 141.4 [92.3 to 216.7] | 443.0 [335.6 to 584.7]

15. Secondary Outcome: Titers for Serum H5N1 HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: as for outcome 1
Time Frame: At Months 6, 12, 18 and 24
Population: The analysis was performed on the ATP cohort for persistence, which consisted of all subjects who had serologic results available at the antibody persistence time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 35 | 40 | 36 | 35 | 46 | 39 | 33 | 40 | 33
Titers
  A/Indonesia/05/2005, Month 6 | 17.6 [10.9 to 28.4] | 17.6 [11.6 to 26.6] | 18.5 [12.1 to 28.5] | 24.3 [16.5 to 35.9] | 17.8 [12.3 to 25.9] | 81.5 [43.4 to 153.0] | 82.5 [47.7 to 142.7] | 42.1 [24.9 to 71.0] | 47.3 [27.5 to 81.5]
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 32 | 39 | 36 | 33 | 44 | 37 | 30 | 39 | 31
  A/Indonesia/05/2005, Month 12 | 19.6 [11.7 to 32.8] | 17.5 [11.3 to 27.2] | 22.4 [15.0 to 33.7] | 19.0 [12.8 to 28.2] | 16.2 [10.9 to 23.9] | 100.2 [53.5 to 187.6] | 108.0 [61.1 to 190.9] | 59.7 [34.8 to 102.3] | 64.7 [37.9 to 110.5]
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 31 | 36 | 29 | 30 | 37 | 34 | 29 | 34 | 29
  A/Indonesia/05/2005, Month 18 | 13.1 [8.2 to 20.8] | 22.9 [15.3 to 34.3] | 20.5 [13.0 to 32.3] | 33.3 [22.1 to 50.3] | 12.0 [8.1 to 18.0] | 55.4 [28.4 to 108.4] | 65.3 [36.0 to 118.3] | 42.5 [25.7 to 70.4] | 55.3 [31.2 to 98.1]
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 30 | 36 | 29 | 27 | 32 | 34 | 28 | 35 | 26
  A/Indonesia/05/2005, Month 24 | 9.9 [6.6 to 14.9] | 9.0 [6.7 to 12.0] | 9.4 [6.5 to 13.6] | 8.7 [6.4 to 11.8] | 10.9 [7.4 to 16.1] | 38.0 [20.1 to 71.8] | 31.2 [16.9 to 57.7] | 21.9 [12.7 to 37.5] | 22.9 [12.9 to 40.4]

16. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroconversion (SCR) was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer < 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strain assessed was Flu A/Indonesia/05/2005.
Time Frame: At Days 7,14, 21, 35 and 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group
Number analyzed (Participants) | 34 | 38 | 33 | 28 | 49
Participants
  A/Indonesia/05/2005, Day 7 | 12 | 17 | 18 | 17 | 0
  A/Indonesia/05/2005, Day 14: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 14 | 22 | 28 | 19 | 21 | 12
  A/Indonesia/05/2005, Day 21: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 21 | 19 | 27 | 19 | 23 | 29
  A/Indonesia/05/2005, Day 35: number analyzed (Participants) | 33 | 36 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 35 | 21 | 33 | 23 | 27 | 49
  A/Indonesia/05/2005, Day 42: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 42 | 22 | 34 | 23 | 27 | 48

17. Secondary Outcome: Number of Seroconverted (SCR) Subjects for HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: SCR was defined as the proportion of subjects who had either a pre-vaccination reciprocal HI titer< 10 and a post-vaccination reciprocal titer ≥ 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post-vaccination reciprocal titer against the vaccine virus. The flu strain assessed was Flu A/Indonesia/05/2005.
Time Frame: At Months 6, 12, 18 and 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 35 | 40 | 36 | 35 | 46 | 38 | 32 | 40 | 32
Participants
  A/Indonesia/05/2005, Month 6 | 12 | 12 | 15 | 14 | 15 | 26 | 24 | 20 | 24
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 32 | 39 | 36 | 33 | 44 | 36 | 29 | 39 | 30
  A/Indonesia/05/2005, Month 12 | 12 | 13 | 17 | 13 | 16 | 27 | 24 | 27 | 23
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 31 | 36 | 29 | 30 | 37 | 33 | 29 | 34 | 28
  A/Indonesia/05/2005, Month 18 | 8 | 17 | 15 | 19 | 5 | 21 | 20 | 22 | 21
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 30 | 36 | 29 | 27 | 32 | 33 | 28 | 35 | 25
  A/Indonesia/05/2005, Month 24 | 7 | 5 | 7 | 3 | 5 | 18 | 16 | 16 | 11

18. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Neutralizing HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroconversion rate for anti-HA antibody response was defined as the percentage of vaccines who have either a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:56 or a pre-vaccination titer ≥ 1:56 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Days 21 (post-vaccination one) and 42 (post-vaccination two)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A AD F1 Primed Group | Control Group
Number analyzed (Participants) | 34 | 38 | 49
Participants
  A/Indonesia/05/2005, Day 21: number analyzed (Participants) | 34 | 0 | 49
  A/Indonesia/05/2005, Day 21 | 29 |  | 44
  A/Indonesia/05/2005, Day 42 | 31 | 35 | 49

19. Secondary Outcome: Number of Seroconverted (SCR) Subjects for Neutralizing HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroconversion rate for neutralizing antibody response was defined as the percentage of vaccines who have either a pre-vaccination titer < 1:40 and a post-vaccination titer ≥ 1:56 or a pre-vaccination titer ≥ 1:56 and at least a 4-fold increase in post-vaccination titer.
Time Frame: At Months 6, 12, 18 and 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A AD F1 Primed Group | Control Group
Number analyzed (Participants) | 37 | 35 | 46
Participants
  A/Indonesia/05/2005, Month 6 | 29 | 29 | 44
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 36 | 32 | 44
  A/Indonesia/05/2005, Month 12 | 17 | 14 | 41
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 33 | 31 | 37
  A/Indonesia/05/2005, Month 18 | 21 | 19 | 35
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 33 | 30 | 32
  A/Indonesia/05/2005, Month 24 | 13 | 13 | 29

20. Secondary Outcome: Seroconversion Factor (SCF) for H5N1 Haemagglutinin-inhibition (HI) Antibodies Against the A/Indonesia/05/2005 Strain
Description: as for outcome 4
Time Frame: At Days 7, 14, 21, 35 and 42
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group
Number analyzed (Participants) | 34 | 38 | 33 | 28 | 49
Fold increase
  A/Indonesia/05/2005, Day 7 | 4.3 [2.3 to 8.2] | 5.1 [2.9 to 8.9] | 5.5 [3.2 to 9.5] | 7.5 [3.9 to 14.7] | 1.0 [1.0 to 1.0]
  A/Indonesia/05/2005, Day 14: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 14 | 9.1 [4.7 to 17.7] | 13.2 [7.9 to 22.0] | 9.8 [5.1 to 18.8] | 14.3 [7.8 to 26.2] | 2.7 [1.9 to 3.9]
  A/Indonesia/05/2005, Day 21: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 21 | 7.4 [4.0 to 13.8] | 11.5 [7.4 to 18.0] | 8.4 [4.6 to 15.5] | 15.4 [9.0 to 26.3] | 6.2 [4.2 to 9.3]
  A/Indonesia/05/2005, Day 35: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 35 | 11.0 [5.6 to 21.4] | 24.0 [15.5 to 37.1] | 13.2 [7.2 to 24.0] | 32.0 [20.2 to 50.8] | 112.7 [87.7 to 144.9]
  A/Indonesia/05/2005, Day 42: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 42 | 10.6 [5.5 to 20.7] | 23.3 [15.4 to 35.1] | 12.7 [6.9 to 23.6] | 28.3 [18.5 to 43.3] | 88.6 [67.1 to 116.9]

21. Secondary Outcome: Seroconversion Factor (SCF) for H5N1 Haemagglutinin-inhibition (HI) Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroconversion factor (SCF) was defined as the fold increase in H5N1 HI antibody GMTs post-vaccination compared to Day 0. The flu strains assessed were A/Indonesia/05/2005.
Time Frame: At Months 6, 12, 18 and 24
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 35 | 40 | 36 | 35 | 46 | 38 | 32 | 40 | 32
Fold increase
  A/Indonesia/05/2005, Month 6 | 3.4 [2.1 to 5.5] | 3.3 [2.3 to 4.8] | 3.7 [2.4 to 5.7] | 4.9 [3.3 to 7.2] | 3.6 [2.5 to 5.2] | 15.0 [8.0 to 28.2] | 14.1 [8.1 to 24.2] | 7.9 [4.8 to 13.1] | 9.8 [5.8 to 16.7]
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 32 | 39 | 36 | 33 | 44 | 36 | 29 | 39 | 30
  A/Indonesia/05/2005, Month 12 | 3.8 [2.3 to 6.4] | 3.3 [2.2 to 4.9] | 4.5 [3.0 to 6.7] | 3.8 [2.6 to 5.6] | 3.2 [2.2 to 4.8] | 18.3 [9.8 to 34.2] | 18.3 [10.4 to 32.1] | 11.2 [6.7 to 18.9] | 13.6 [8.1 to 22.8]
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 31 | 36 | 29 | 30 | 37 | 33 | 29 | 34 | 28
  A/Indonesia/05/2005, Month 18 | 2.6 [1.6 to 4.0] | 4.6 [3.1 to 6.9] | 4.1 [2.6 to 6.5] | 6.7 [4.4 to 10.1] | 2.4 [1.6 to 3.6] | 10.1 [5.2 to 19.7] | 11.5 [6.5 to 20.3] | 7.9 [4.9 to 12.8] | 11.6 [6.7 to 20.2]
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 30 | 36 | 29 | 27 | 32 | 33 | 28 | 35 | 25
  A/Indonesia/05/2005, Month 24 | 1.9 [1.3 to 2.9] | 1.8 [1.3 to 2.4] | 1.9 [1.3 to 2.7] | 1.7 [1.3 to 2.4] | 2.2 [1.5 to 3.2] | 6.9 [3.7 to 13.0] | 5.9 [3.2 to 10.7] | 4.1 [2.4 to 6.8] | 4.7 [2.6 to 8.3]

22. Secondary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: Seroprotection rate was defined as the percentage of vaccines with a serum HI antibody titer ≥ 1:40 that usually is accepted as indicating protection.
  The flu strain assessed was A/Indonesia/05/2005 (H5N1).
Time Frame: At Days 0, 7, 14, 21, 28, 35 and 42
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group
Number analyzed (Participants) | 34 | 38 | 33 | 28 | 49
Participants
  A/Indonesia/05/2005, Day 0 | 0 | 0 | 0 | 0 | 0
  A/Indonesia/05/2005, Day 7: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 7 | 12 | 17 | 18 | 17 | 0
  A/Indonesia/05/2005, Day 14: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 14 | 22 | 28 | 19 | 21 | 12
  A/Indonesia/05/2005, Day 21: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 21 | 19 | 27 | 19 | 23 | 29
  A/Indonesia/05/2005, Day 28: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 28 | 22 | 32 | 22 | 26 | 49
  A/Indonesia/05/2005, Day 35: number analyzed (Participants) | 33 | 36 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 35 | 21 | 33 | 23 | 27 | 49
  A/Indonesia/05/2005, Day 42: number analyzed (Participants) | 34 | 38 | 32 | 28 | 49
  A/Indonesia/05/2005, Day 42 | 22 | 34 | 23 | 27 | 48

23. Secondary Outcome: Number of Seroprotected (SPR) Subjects for HI Antibodies Against the A/Indonesia/05/2005 Strain
Description: as for outcome 22
Time Frame: At Months 6, 12, 18 and 24
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
Number analyzed (Participants) | 35 | 40 | 36 | 35 | 46 | 39 | 33 | 40 | 33
Participants
  A/Indonesia/05/2005, Month 6 | 12 | 12 | 15 | 14 | 15 | 27 | 25 | 20 | 24
  A/Indonesia/05/2005, Month 12: number analyzed (Participants) | 32 | 39 | 36 | 33 | 44 | 37 | 30 | 39 | 31
  A/Indonesia/05/2005, Month 12 | 12 | 13 | 17 | 13 | 16 | 28 | 25 | 27 | 23
  A/Indonesia/05/2005, Month 18: number analyzed (Participants) | 31 | 36 | 29 | 30 | 37 | 34 | 29 | 34 | 29
  A/Indonesia/05/2005, Month 18 | 8 | 17 | 15 | 19 | 5 | 22 | 20 | 22 | 21
  A/Indonesia/05/2005, Month 24: number analyzed (Participants) | 30 | 36 | 29 | 27 | 32 | 34 | 28 | 35 | 26
  A/Indonesia/05/2005, Month 24 | 7 | 5 | 7 | 3 | 5 | 19 | 16 | 16 | 11

24. Secondary Outcome: Frequency of Antigen-specific CD4/CD8 T-cells (Per 10E6) in Tests Identified as Producing at Least Two Out of Four Different Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 4 all doubles (CD4 all doubles), cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). The flu strains assessed wwere H5N1 A/Indonesia and H5N1 A/Vietnam.
Time Frame: At Days 0 and 21
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: T-cells/million cells
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A AD F1 Primed Group | Control Group
Number analyzed (Participants) | 32 | 38 | 48
T-cells/million cells
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Day 0 | 743.00 [524.00 to 991.00] | 1370.00 [776.00 to 1599.00] | 473.50 [277.50 to 757.00]
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Day 21 | 1945.50 [1104.50 to 2737.50] | 2504.00 [1515.00 to 4252.00] | 2721.00 [2040.00 to 4072.00]
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Day 0 | 682.50 [475.00 to 1044.50] | 1284.50 [839.00 to 1831.00] | 540.00 [379.00 to 873.50]
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Day 21 | 1870.00 [1179.50 to 2806.50] | 2640.50 [1217.00 to 4211.00] | 2607.00 [1973.00 to 3738.00]
  CD4 CD40L - H5N1 A/Indonesia, Day 0 | 709.00 [484.50 to 1014.00] | 1363.50 [721.00 to 1546.00] | 457.50 [280.50 to 738.00]
  CD4 CD40L - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 CD40L - H5N1 A/Indonesia, Day 21 | 1874.00 [1093.50 to 2657.50] | 2480.00 [1501.00 to 3972.00] | 2633.00 [1894.00 to 4033.00]
  CD4 CD40L - H5N1 A/Vietnam, Day 0 | 650.00 [470.50 to 1011.00] | 1288.50 [832.00 to 1830.00] | 525.50 [366.00 to 832.50]
  CD4 CD40L - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 CD40L - H5N1 A/Vietnam, Day 21 | 1842.50 [1145.50 to 2727.00] | 2652.00 [1218.00 to 4039.00] | 2580.50 [1847.00 to 3578.00]
  CD4 IL-2 - H5N1 A/Indonesia, Day 0 | 641.00 [419.50 to 847.00] | 1186.50 [773.00 to 1492.00] | 433.50 [273.50 to 671.00]
  CD4 IL-2 - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 IL-2 - H5N1 A/Indonesia, Day 21 | 1616.00 [1044.00 to 2475.00] | 2291.50 [1474.00 to 3648.00] | 2485.00 [1800.00 to 3839.00]
  CD4 IL-2 - H5N1 A/Vietnam, Day 0 | 599.50 [381.50 to 931.50] | 1195.50 [744.00 to 1635.00] | 473.50 [339.00 to 778.50]
  CD4 IL-2 - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 IL-2 - H5N1 A/Vietnam, Day 21 | 1607.00 [1064.00 to 2588.50] | 2210.00 [1120.00 to 3828.00] | 2368.50 [1840.00 to 3458.00]
  CD4 INF-γ - H5N1 A/Indonesia, Day 0 | 407.00 [282.00 to 626.00] | 607.00 [388.00 to 873.00] | 357.00 [203.50 to 518.50]
  CD4 INF-γ - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 INF-γ - H5N1 A/Indonesia, Day 21 | 785.50 [472.00 to 1453.00] | 1304.50 [613.00 to 1829.00] | 993.50 [735.00 to 1840.00]
  CD4 INF-γ - H5N1 A/Vietnam, Day 0 | 470.00 [233.50 to 731.00] | 729.50 [440.00 to 1012.00] | 406.50 [282.00 to 685.50]
  CD4 INF-γ - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 INF-γ - H5N1 A/Vietnam, Day 21 | 960.50 [604.50 to 1568.00] | 1105.00 [662.00 to 1958.00] | 1057.50 [855.00 to 1707.00]
  CD4 TNF-α - H5N1 A/Indonesia, Day 0 | 544.00 [405.00 to 708.50] | 944.50 [652.00 to 1219.00] | 294.00 [173.00 to 509.50]
  CD4 TNF-α - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 TNF-α - H5N1 A/Indonesia, Day 21 | 1187.00 [729.00 to 1882.00] | 1905.50 [1019.00 to 2972.00] | 1658.50 [1093.00 to 2342.00]
  CD4 TNF-α - H5N1 A/Vietnam, Day 0 | 490.50 [364.50 to 772.50] | 952.50 [665.00 to 1406.00] | 357.00 [232.50 to 692.50]
  CD4 TNF-α - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD4 TNF-α - H5N1 A/Vietnam, Day 21 | 1360.00 [709.00 to 1925.50] | 1888.00 [894.00 to 3102.00] | 1616.50 [1307.00 to 2160.00]
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Day 0 | 71.00 [10.00 to 205.00] | 60.50 [3.00 to 256.00] | 47.50 [1.00 to 170.50]
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Day 21 | 132.50 [30.00 to 251.00] | 75.00 [1.00 to 258.00] | 52.00 [25.00 to 143.00]
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Day 0 | 159.00 [43.50 to 425.00] | 99.50 [37.00 to 244.00] | 90.50 [2.00 to 343.50]
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Day 21 | 166.50 [93.50 to 463.00] | 153.00 [42.00 to 316.00] | 147.50 [58.00 to 357.00]
  CD8 CD40L - H5N1 A/Indonesia, Day 0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  CD8 CD40L - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 CD40L - H5N1 A/Indonesia, Day 21 | 1.00 [1.00 to 11.50] | 1.00 [1.00 to 13.00] | 1.00 [1.00 to 1.00]
  CD8 CD40L - H5N1 A/Vietnam, Day 0 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 25.00] | 1.00 [1.00 to 1.00]
  CD8 CD40L - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 CD40L - H5N1 A/Vietnam, Day 21 | 1.00 [1.00 to 32.50] | 1.00 [1.00 to 27.00] | 1.00 [1.00 to 1.00]
  CD8 IL-2 - H5N1 A/Indonesia, Day 0 | 42.50 [1.00 to 116.50] | 40.00 [1.00 to 190.00] | 30.50 [1.00 to 113.00]
  CD8 IL-2 - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 IL-2 - H5N1 A/Indonesia, Day 21 | 31.00 [1.00 to 142.50] | 39.00 [1.00 to 167.00] | 39.00 [1.00 to 90.00]
  CD8 IL-2 - H5N1 A/Vietnam, Day 0 | 59.50 [24.50 to 150.00] | 48.50 [22.00 to 178.00] | 51.00 [1.00 to 183.00]
  CD8 IL-2 - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 IL-2 - H5N1 A/Vietnam, Day 21 | 86.00 [39.00 to 203.50] | 90.50 [29.00 to 162.00] | 86.50 [31.00 to 219.00]
  CD8 INF-γ - H5N1 A/Indonesia, Day 0 | 92.00 [1.00 to 218.50] | 40.50 [1.00 to 207.00] | 37.50 [1.00 to 155.00]
  CD8 INF-γ - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 INF-γ - H5N1 A/Indonesia, Day 21 | 132.50 [31.00 to 261.50] | 56.50 [1.00 to 255.00] | 41.00 [4.00 to 136.00]
  CD8 INF-γ - H5N1 A/Vietnam, Day 0 | 152.50 [27.00 to 425.00] | 76.00 [35.00 to 223.00] | 97.50 [16.50 to 342.50]
  CD8 INF-γ - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 INF-γ - H5N1 A/Vietnam, Day 21 | 150.00 [82.50 to 444.00] | 127.00 [38.00 to 287.00] | 149.00 [58.00 to 350.00]
  CD8 TNF-α - H5N1 A/Indonesia, Day 0 | 80.00 [1.00 to 177.50] | 47.00 [1.00 to 161.00] | 28.00 [1.00 to 138.50]
  CD8 TNF-α - H5N1 A/Indonesia, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 TNF-α - H5N1 A/Indonesia, Day 21 | 124.50 [26.00 to 239.00] | 75.50 [1.00 to 162.00] | 36.50 [1.00 to 89.00]
  CD8 TNF-α - H5N1 A/Vietnam, Day 0 | 98.50 [18.50 to 425.00] | 83.00 [25.00 to 178.00] | 71.00 [1.00 to 208.50]
  CD8 TNF-α - H5N1 A/Vietnam, Day 21: number analyzed (Participants) | 32 | 38 | 46
  CD8 TNF-α - H5N1 A/Vietnam, Day 21 | 115.00 [41.50 to 429.00] | 98.00 [32.00 to 246.00] | 136.00 [1.00 to 350.00]

25. Secondary Outcome: Frequency of Antigen-specific CD4/CD8 T-cells (Per 10E6) in Tests Identified as Producing at Least Two Out of Four Different Cytokines
Description: Among cytokines expressed after background reduction were cluster of differentiation 4 all doubles (CD4 all doubles), cluster of differentiation 40-ligand (CD40-L), interleukin-2 (IL-2), interferon-gamma (IFN-γ) and tumour necrosis factor-alpha (TNF-α). The flu strains assessed were H5N1 A/Indonesia and H5N1 A/Vietnam.
Time Frame: At Months 6, 12, 18 and 24
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: T-cell/million cells
Arm/Group | GSK1562902A AD F1 Primed Group | GSK1562902A Non-AD F1 Primed Group | Control Group
Number analyzed (Participants) | 37 | 35 | 45
T-cell/million cells
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 6 | 1575.00 [1157.00 to 2247.00] | 1244.00 [919.00 to 1816.00] | 1817.00 [1296.00 to 2235.00]
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 6 | 1710.00 [1063.00 to 2393.00] | 1138.00 [929.00 to 1677.00] | 1775.00 [1208.00 to 2156.00]
  CD4 CD40L - H5N1 A/Indonesia, Month 6 | 1605.00 [1157.00 to 2199.00] | 1190.00 [903.00 to 1734.00] | 1720.00 [1202.00 to 2188.00]
  CD4 CD40L - H5N1 A/Vietnam, Month 6 | 1724.00 [1049.00 to 2281.00] | 1124.00 [890.00 to 1636.00] | 1748.00 [1140.00 to 2169.00]
  CD4 IL-2 - H5N1 A/Indonesia, Month 6 | 1454.00 [1031.00 to 2111.00] | 1136.00 [780.00 to 1683.00] | 1736.00 [1140.00 to 2122.00]
  CD4 IL-2 - H5N1 A/Vietnam, Month 6 | 1481.00 [979.00 to 2183.00] | 1070.00 [782.00 to 1555.00] | 1580.00 [1070.00 to 2023.00]
  CD4 INF-γ - H5N1 A/Indonesia, Month 6 | 794.00 [516.00 to 1228.00] | 636.00 [411.00 to 1015.00] | 929.00 [571.00 to 1235.00]
  CD4 INF-γ - H5N1 A/Vietnam, Month 6 | 876.00 [547.00 to 1376.00] | 679.00 [413.00 to 914.00] | 885.00 [599.00 to 1284.00]
  CD4 TNF-α - H5N1 A/Indonesia, Month 6 | 1152.00 [848.00 to 1836.00] | 920.00 [698.00 to 1322.00] | 1467.00 [1004.00 to 1890.00]
  CD4 TNF-α - H5N1 A/Vietnam, Month 6 | 1279.00 [860.00 to 1984.00] | 941.00 [716.00 to 1169.00] | 1292.00 [936.00 to 1771.00]
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 12 | 1333.00 [903.00 to 1981.00] | 786.50 [560.50 to 1074.50] | 1332.50 [846.00 to 1566.00]
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 12 | 1171.00 [813.00 to 1851.00] | 796.50 [591.50 to 1148.50] | 1225.00 [786.00 to 1565.50]
  CD4 CD40L - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 CD40L - H5N1 A/Indonesia, Month 12 | 1119.00 [580.00 to 1604.00] | 647.00 [406.50 to 938.50] | 1159.00 [746.00 to 1472.50]
  CD4 CD40L - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 CD40L - H5N1 A/Vietnam, Month 12 | 1090.00 [728.00 to 1632.00] | 641.00 [395.50 to 947.00] | 1134.00 [679.50 to 1355.50]
  CD4 IL-2 - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 IL-2 - H5N1 A/Indonesia, Month 12 | 1290.00 [860.00 to 1826.00] | 721.00 [490.50 to 1038.00] | 1219.50 [805.00 to 1525.50]
  CD4 IL-2 - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 IL-2 - H5N1 A/Vietnam, Month 12 | 1183.00 [746.00 to 1842.00] | 733.00 [540.00 to 1055.00] | 1100.00 [745.00 to 1466.00]
  CD4 INF-γ - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 INF-γ - H5N1 A/Indonesia, Month 12 | 746.00 [485.00 to 958.00] | 432.50 [346.00 to 657.50] | 618.00 [382.50 to 839.50]
  CD4 INF-γ - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 INF-γ - H5N1 A/Vietnam, Month 12 | 670.00 [512.00 to 1033.00] | 497.50 [299.00 to 679.50] | 643.00 [372.50 to 979.50]
  CD4 TNF-α - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 TNF-α - H5N1 A/Indonesia, Month 12 | 1065.00 [692.00 to 1623.00] | 551.50 [432.00 to 814.50] | 997.50 [665.50 to 1272.50]
  CD4 TNF-α - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD4 TNF-α - H5N1 A/Vietnam, Month 12 | 945.00 [728.00 to 1534.00] | 616.50 [474.50 to 796.00] | 939.50 [620.00 to 1226.50]
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 18 | 1421.00 [959.00 to 2106.00] | 1052.00 [748.00 to 1705.00] | 1392.00 [1119.00 to 2003.00]
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 18 | 1536.00 [893.00 to 2061.00] | 1022.00 [699.00 to 1665.00] | 1367.00 [995.00 to 1650.00]
  CD4 CD40L - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 CD40L - H5N1 A/Indonesia, Month 18 | 1369.00 [869.00 to 2080.00] | 1013.00 [733.00 to 1679.00] | 1330.00 [1083.00 to 1937.00]
  CD4 CD40L - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 CD40L - H5N1 A/Vietnam, Month 18 | 1523.00 [821.00 to 2088.00] | 1036.00 [634.00 to 1653.00] | 1288.00 [997.00 to 1642.00]
  CD4 IL-2 - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 IL-2 - H5N1 A/Indonesia, Month 18 | 1316.00 [829.00 to 1868.00] | 946.00 [613.00 to 1434.00] | 1170.00 [929.00 to 1511.00]
  CD4 IL-2 - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 IL-2 - H5N1 A/Vietnam, Month 18 | 1346.00 [817.00 to 1942.00] | 933.00 [578.00 to 1354.00] | 1062.00 [925.00 to 1475.00]
  CD4 INF-γ - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 INF-γ - H5N1 A/Indonesia, Month 18 | 906.00 [553.00 to 1592.00] | 729.00 [490.00 to 1158.00] | 865.00 [655.00 to 1424.00]
  CD4 INF-γ - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 INF-γ - H5N1 A/Vietnam, Month 18 | 1042.00 [560.00 to 1519.00] | 743.00 [523.00 to 1292.00] | 965.00 [670.00 to 1343.00]
  CD4 TNF-α - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 TNF-α - H5N1 A/Indonesia, Month 18 | 1173.00 [764.00 to 1600.00] | 811.00 [577.00 to 1142.00] | 1035.00 [824.00 to 1490.00]
  CD4 TNF-α - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD4 TNF-α - H5N1 A/Vietnam, Month 18 | 1074.00 [693.00 to 1623.00] | 793.00 [563.00 to 1195.00] | 1079.00 [748.00 to 1431.00]
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 ALL DOUBLES - H5N1 A/Indonesia, Month 24 | 1307.00 [946.00 to 1588.00] | 914.00 [759.00 to 1381.00] | 1306.00 [795.00 to 1632.00]
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 ALL DOUBLES - H5N1 A/Vietnam, Month 24 | 1229.00 [872.00 to 1746.00] | 850.00 [565.00 to 1327.00] | 1322.00 [877.00 to 1606.00]
  CD4 CD40L - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 CD40L - H5N1 A/Indonesia, Month 24 | 1220.00 [893.00 to 1585.00] | 917.00 [745.00 to 1237.00] | 1280.00 [739.00 to 1580.00]
  CD4 CD40L - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 CD40L - H5N1 A/Vietnam, Month 24 | 1195.00 [885.00 to 1733.00] | 826.00 [565.00 to 1314.00] | 1356.00 [851.00 to 1576.00]
  CD4 IL-2 - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 IL-2 - H5N1 A/Indonesia, Month 24 | 1146.00 [796.00 to 1402.00] | 867.00 [692.00 to 1139.00] | 1105.00 [646.00 to 1460.00]
  CD4 IL-2 - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 IL-2 - H5N1 A/Vietnam, Month 24 | 1101.00 [787.00 to 1533.00] | 839.00 [493.00 to 1211.00] | 1253.00 [686.00 to 1369.00]
  CD4 INF-γ - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 INF-γ - H5N1 A/Indonesia, Month 24 | 848.00 [597.00 to 1124.00] | 654.00 [492.00 to 975.00] | 860.00 [458.00 to 1087.00]
  CD4 INF-γ - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 INF-γ - H5N1 A/Vietnam, Month 24 | 838.00 [517.00 to 1031.00] | 704.00 [464.00 to 991.00] | 888.00 [512.00 to 1130.00]
  CD4 TNF-α - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 TNF-α - H5N1 A/Indonesia, Month 24 | 1062.00 [730.00 to 1306.00] | 773.00 [654.00 to 965.00] | 1186.00 [627.00 to 1437.00]
  CD4 TNF-α - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD4 TNF-α - H5N1 A/Vietnam, Month 24 | 999.00 [770.00 to 1253.00] | 680.00 [441.00 to 1085.00] | 1023.00 [593.00 to 1329.00]
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 6 | 59.00 [1.00 to 184.00] | 79.00 [16.00 to 264.00] | 89.00 [1.00 to 199.00]
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 6 | 85.00 [53.00 to 288.00] | 139.00 [61.00 to 286.00] | 107.00 [1.00 to 241.00]
  CD8 CD40L - H5N1 A/Indonesia, Month 6 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 23.00] | 1.00 [1.00 to 1.00]
  CD8 CD40L - H5N1 A/Vietnam, Month 6 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  CD8 IL-2 - H5N1 A/Indonesia, Month 6 | 52.00 [1.00 to 107.00] | 54.00 [1.00 to 240.00] | 53.00 [1.00 to 115.00]
  CD8 IL-2 - H5N1 A/Vietnam, Month 6 | 93.00 [18.00 to 227.00] | 77.00 [27.00 to 182.00] | 63.00 [1.00 to 158.00]
  CD8 INF-γ - H5N1 A/Indonesia, Month 6 | 29.00 [1.00 to 158.00] | 49.00 [1.00 to 202.00] | 44.00 [1.00 to 165.00]
  CD8 INF-γ - H5N1 A/Vietnam, Month 6 | 48.00 [1.00 to 239.00] | 117.00 [21.00 to 246.00] | 61.00 [1.00 to 221.00]
  CD8 TNF-α - H5N1 A/Indonesia, Month 6 | 52.00 [1.00 to 99.00] | 71.00 [1.00 to 216.00] | 76.00 [1.00 to 146.00]
  CD8 TNF-α - H5N1 A/Vietnam, Month 6 | 73.00 [18.00 to 218.00] | 123.00 [59.00 to 246.00] | 80.00 [1.00 to 215.00]
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 12 | 78.00 [26.00 to 166.00] | 73.00 [3.00 to 172.00] | 30.50 [1.00 to 94.50]
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 12 | 69.00 [21.00 to 210.00] | 95.00 [17.00 to 293.00] | 31.50 [1.00 to 104.50]
  CD8 CD40L - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 CD40L - H5N1 A/Indonesia, Month 12 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  CD8 CD40L - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 CD40L - H5N1 A/Vietnam, Month 12 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 1.00]
  CD8 IL-2 - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 IL-2 - H5N1 A/Indonesia, Month 12 | 56.00 [2.00 to 166.00] | 54.50 [1.00 to 117.50] | 5.50 [1.00 to 82.50]
  CD8 IL-2 - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 IL-2 - H5N1 A/Vietnam, Month 12 | 55.00 [1.00 to 142.00] | 49.50 [2.00 to 186.00] | 13.00 [1.00 to 78.00]
  CD8 INF-γ - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 INF-γ - H5N1 A/Indonesia, Month 12 | 46.00 [1.00 to 168.00] | 60.50 [1.00 to 159.50] | 1.00 [1.00 to 80.50]
  CD8 INF-γ - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 INF-γ - H5N1 A/Vietnam, Month 12 | 77.00 [31.00 to 205.00] | 54.00 [13.00 to 263.50] | 32.00 [1.00 to 131.00]
  CD8 TNF-α - H5N1 A/Indonesia, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 TNF-α - H5N1 A/Indonesia, Month 12 | 54.00 [11.00 to 109.00] | 62.00 [1.00 to 117.50] | 23.50 [1.00 to 66.50]
  CD8 TNF-α - H5N1 A/Vietnam, Month 12: number analyzed (Participants) | 37 | 28 | 44
  CD8 TNF-α - H5N1 A/Vietnam, Month 12 | 55.00 [1.00 to 158.00] | 75.50 [7.00 to 224.00] | 31.50 [1.00 to 92.00]
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 18 | 35.00 [1.00 to 208.00] | 82.00 [1.00 to 160.00] | 40.00 [1.00 to 127.00]
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 18 | 48.00 [1.00 to 138.00] | 66.00 [28.00 to 214.00] | 119.00 [28.00 to 270.00]
  CD8 CD40L - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 CD40L - H5N1 A/Indonesia, Month 18 | 1.00 [1.00 to 29.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 30.00]
  CD8 CD40L - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 CD40L - H5N1 A/Vietnam, Month 18 | 1.00 [1.00 to 64.00] | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 75.00]
  CD8 IL-2 - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 IL-2 - H5N1 A/Indonesia, Month 18 | 1.00 [1.00 to 68.00] | 43.00 [1.00 to 99.00] | 30.00 [1.00 to 90.00]
  CD8 IL-2 - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 IL-2 - H5N1 A/Vietnam, Month 18 | 1.00 [1.00 to 98.00] | 40.00 [1.00 to 170.00] | 47.00 [1.00 to 79.00]
  CD8 TNF-α - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 TNF-α - H5N1 A/Indonesia, Month 18 | 38.00 [1.00 to 177.00] | 82.00 [1.00 to 162.00] | 31.00 [1.00 to 127.00]
  CD8 INF-γ - H5N1 A/Indonesia, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 INF-γ - H5N1 A/Indonesia, Month 18 | 48.00 [1.00 to 138.00] | 62.00 [9.00 to 214.00] | 119.00 [24.00 to 270.00]
  CD8 INF-γ - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 INF-γ - H5N1 A/Vietnam, Month 18 | 1.00 [1.00 to 157.00] | 81.00 [1.00 to 205.00] | 42.00 [1.00 to 109.00]
  CD8 TNF-α - H5N1 A/Vietnam, Month 18: number analyzed (Participants) | 33 | 31 | 37
  CD8 TNF-α - H5N1 A/Vietnam, Month 18 | 38.00 [1.00 to 132.00] | 65.00 [22.00 to 240.00] | 107.00 [30.00 to 158.00]
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 ALL DOUBLES - H5N1 A/Indonesia, Month 24 | 78.00 [1.00 to 167.00] | 73.00 [1.00 to 247.00] | 65.00 [1.00 to 148.00]
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 ALL DOUBLES - H5N1 A/Vietnam, Month 24 | 29.00 [1.00 to 243.00] | 73.00 [1.00 to 193.00] | 102.00 [1.00 to 269.00]
  CD8 CD40L - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 CD40L - H5N1 A/Indonesia, Month 24 | 26.00 [1.00 to 65.00] | 1.00 [1.00 to 36.00] | 1.00 [1.00 to 44.00]
  CD8 CD40L - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 CD40L - H5N1 A/Vietnam, Month 24 | 1.00 [1.00 to 47.00] | 1.00 [1.00 to 44.00] | 1.00 [1.00 to 93.00]
  CD8 IL-2 - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 IL-2 - H5N1 A/Indonesia, Month 24 | 21.00 [1.00 to 62.00] | 25.00 [1.00 to 115.00] | 32.00 [1.00 to 68.00]
  CD8 IL-2 - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 IL-2 - H5N1 A/Vietnam, Month 24 | 1.00 [1.00 to 77.00] | 26.00 [1.00 to 99.00] | 31.00 [1.00 to 130.00]
  CD8 INF-γ - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 INF-γ - H5N1 A/Indonesia, Month 24 | 64.00 [1.00 to 167.00] | 93.00 [1.00 to 231.00] | 65.00 [1.00 to 143.00]
  CD8 INF-γ - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 INF-γ - H5N1 A/Vietnam, Month 24 | 31.00 [1.00 to 243.00] | 73.00 [1.00 to 193.00] | 102.00 [22.00 to 231.00]
  CD8 TNF-α - H5N1 A/Indonesia, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 TNF-α - H5N1 A/Indonesia, Month 24 | 26.00 [1.00 to 128.00] | 57.00 [1.00 to 153.00] | 55.00 [1.00 to 89.00]
  CD8 TNF-α - H5N1 A/Vietnam, Month 24: number analyzed (Participants) | 33 | 31 | 37
  CD8 TNF-α - H5N1 A/Vietnam, Month 24 | 37.00 [1.00 to 174.00] | 45.00 [1.00 to 148.00] | 64.00 [1.00 to 182.00]

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events (AEs): during the 21-day (Days 0-20) or 30-day (Days 0-29) post-vaccination 1 period and the 30-day (Days 0-29) post-vaccination 2 period; Serious adverse events (SAEs): during the whole study period (from Day 0 up to Month 24).
Arm/Group | GSK1562902A Non-AD F1 Primed Group | GSK1562902A Non-AD F2 Primed Group | GSK1562902A Non-AD F3 Primed Group | GSK1562902A Non-AD F4 Primed Group | Control Group | GSK1562902A AD F1 Primed Group | GSK1562902A AD F2 Primed Group | GSK1562902A AD F3 Primed Group | GSK1562902A AD Approved F Primed Group
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/40 | 0/37 | 0/36 | 0/50 | 0/40 | 0/35 | 1/41 | 1/35
Serious Adverse Events (participants affected / at risk) | 4/36 | 3/40 | 2/37 | 0/36 | 4/50 | 2/40 | 1/35 | 4/41 | 3/35
Other Adverse Events (participants affected / at risk) | 34/36 | 40/40 | 33/37 | 35/36 | 48/50 | 39/40 | 34/35 | 41/41 | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A Non-AD F1 Primed Group (N=36) | GSK1562902A Non-AD F2 Primed Group (N=40) | GSK1562902A Non-AD F3 Primed Group (N=37) | GSK1562902A Non-AD F4 Primed Group (N=36) | Control Group (N=50) | GSK1562902A AD F1 Primed Group (N=40) | GSK1562902A AD F2 Primed Group (N=35) | GSK1562902A AD F3 Primed Group (N=41) | GSK1562902A AD Approved F Primed Group (N=35)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ill-defined disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Traumatic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
High grade b-cell lymphoma burkitt-like lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Major depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic aneurysm rupture (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSK1562902A Non-AD F1 Primed Group (N=36) | GSK1562902A Non-AD F2 Primed Group (N=40) | GSK1562902A Non-AD F3 Primed Group (N=37) | GSK1562902A Non-AD F4 Primed Group (N=36) | Control Group (N=50) | GSK1562902A AD F1 Primed Group (N=40) | GSK1562902A AD F2 Primed Group (N=35) | GSK1562902A AD F3 Primed Group (N=41) | GSK1562902A AD Approved F Primed Group (N=35)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (16) | 8 (11) | 6 (7) | 11 (12) | 15 (20) | 6 (7) | 5 (5) | 5 (5) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 10 (11) | 3 (4) | 4 (5) | 7 (8) | 20 (21) | 9 (9) | 6 (6) | 6 (7) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 4 (6) | 2 (2) | 2 (3) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (3) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Fatigue (General disorders) | 20 (25) | 22 (28) | 18 (25) | 20 (28) | 30 (51) | 15 (16) | 10 (11) | 18 (19) | 14 (14)
Headache (Nervous system disorders) | 22 (33) | 19 (30) | 18 (32) | 18 (30) | 31 (49) | 19 (23) | 12 (13) | 13 (15) | 11 (14)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 9 (9) | 4 (6) | 6 (9) | 5 (5) | 13 (20) | 5 (5) | 6 (6) | 4 (5) | 3 (3)
Induration (General disorders) | 6 (6) | 5 (6) | 5 (6) | 2 (3) | 6 (6) | 2 (2) | 4 (4) | 3 (3) | 4 (4)
Influenza like illness (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Injection site reaction (General disorders) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (24) | 21 (27) | 15 (23) | 15 (19) | 30 (42) | 12 (12) | 12 (12) | 11 (12) | 10 (10)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 3 (5) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 3 (4) | 2 (2) | 7 (8) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Pain (General disorders) | 34 (61) | 36 (65) | 32 (56) | 35 (62) | 47 (87) | 38 (38) | 34 (35) | 39 (40) | 31 (32)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 2 (2) | 5 (6) | 0 (0) | 1 (1) | 2 (2) | 6 (6)
Swelling (General disorders) | 5 (7) | 2 (2) | 5 (6) | 6 (9) | 6 (8) | 2 (2) | 3 (3) | 3 (3) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 3 (3) | 3 (3) | 8 (9) | 5 (5) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.